CLINICAL TRIAL: NCT01267318
Title: Evaluation of Gastric Juice Samples During Standard Gastroscopy Procedure
Status: Terminated | Type: Observational
Why Stopped: Sponsor decided to terminate the entire project, and therefore there was no use for the samples collected in the study.
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: RD-301
Record Dates: First submitted 2010-12-26; First posted 2010-12-28 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2012-07

CONDITIONS: Gastrointestinal Bleeding
Keywords: Gastric juice; Stomach; GI; Gastric juice samples with presence of blood.
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gastric juices content suctioned from patients routinely during the course of Gastroscopy.
Oversight: Data Monitoring Committee: No

SUMMARY:
Development of a new diagnostic detection tool for gastrointestinal bleeding.

DETAILED DESCRIPTION:
Literature does not support enough data/knowledge regarding stomach bleeding Hb levels in pathological situations and/or stomach bleeding levels following biopsy. It is important to understand the approximate concentration level of stomach bleeding before proceeding with technology development to insure this technology is capable of detecting such blood levels.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 18 years old.
* Subject is scheduled for EGD endoscopy which includes biopsy, or,
* Subject is scheduled for EGD endoscopy following a bleeding event.

Exclusion Criteria:

* Subject is either not competent or not willing to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All gastric juice samples should contain blood. This will be determined by the treating physician based on visual assessment in a region alongside the fresh biopsy site just performed, and prior to any saline washing.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rami Eliakim, Prof., Principal Investigator — Rambam Health Care Campus
Locations (1):
- RAMBAM Medical Center, Haifa, Israel